CLINICAL TRIAL: NCT05872152
Title: Impact of Fourier Transform Infrared Spectroscopy (FTIRS) on the Diffusion of ESBL Producing Enterobacterales in Intensive Care Units (ICU)
Brief Title: Impact of Fourier Transform Infrared Spectroscopy (FTIRS) in ICUs
Acronym: ECLA'IR
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Caen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Prevention
Other Study IDs: 220145
Record Dates: First submitted 2023-04-11; First posted 2023-05-24 (Actual); Last update posted 2025-07-24 (Actual); Status verified 2025-07

CONDITIONS: Organ Failure, Multiple
Keywords: multidrug resistant bacteria; outbreak; prevention and infection control; bacterial typing; Fourier transform infrared spectroscopy
MeSH Terms: conditions — Multiple Organ Failure

STUDY DESIGN:
Intervention Model Description: Stepped-wedge
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard care (No Intervention): Standard care are defined by routine procedures implemented in each center to prevent and control the diffusion of MDR-E bacteria in ICUs. In the first period of the study, the frequency of cross transmission will be assessed by sequencing the first ESBL-E isolate in each carrier patients (first isolate of a given species)
- Transmission of FTIR results (Experimental): In second phase of the study, the result of FTIR typing of recovered ESBL-E isolates will be weekly transmitted to participating centers.
  Interventions: Diagnostic Test: FTIR results

INTERVENTIONS:
Diagnostic Test: FTIR results — Weekly transmission of FTIRS typing of ESBL-E to centers
  Arms: Transmission of FTIR results

SUMMARY:
This study will assess the impact of FTIRS typing on the spread of ESBL-E in intensive care units

DETAILED DESCRIPTION:
Multidrug resistant enterobacterales (MDR-E) are a major threat for patients hospitalized in intensive care units (ICUs). To prevent MDR-E spread in ICUs, rectal swabs are routinely performed and cultured on selective media. However, bacterial identification and antimicrobial susceptibility results are not sufficient to diagnose cross transmissions. The gold standard technique is based on genomic analysis that require whole genome sequencing (WGS) of bacteria and followed by multilocus sequence typing (MLST) and Single Nucleotide Polymorphism (SNP) typing. This technology is rather expensive and not applicable in all centers.

Fourier Transform InfraRed Spectroscopy (FTIRS) is a developing method for rapid bacterial typing. This technology is simple and results can be obtained in one hour. It is therefore adapted to continuous surveillance of MDR-E. In France, extended spectrum betalactamase producing enterobacteriaceae (ESBL-E) represent the vast majority of MDR-E. We postulate that early diagnosis of cross-transmission by FTIRS may prevent the spread of ESBL-E in ICUs and favor compliance with hygiene measures. The aim of this study will be to assess the impact of systematic FTIRS typing of ESBL-E on ESBL-E cross-transmissions in ICUs.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients hospitalized in ICU
* ESBL-E carrier

Exclusion Criteria:

* none

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 900 (Estimated)
Dates: Start 2024-01-08 (Actual); Primary Completion 2026-09-01 (Estimated); Study Completion 2026-09-01 (Estimated)

PRIMARY OUTCOMES:
Baseline frequency of ESBL-E cross transmission as assessed by WGS | Month 9 to Month 12 (depending on centers, stepped wedge design)
  Number of patients with hospital acquired ESBL-E / total number of ESBL-E carriers
Post intervention frequency of ESBL-E cross transmission as assessed by WGS | Month 24
  Number of patients with hospital acquired ESBL-E / total number of ESBL-E carriers

SECONDARY OUTCOMES:
Sensitivity of FTIRS to diagnose cross transmissions compared to WGS | Month 24
  Sensitivity
Specificity of FTIRS to diagnose cross transmissions compared to WGS | Month 24
  Specificity
Positive predictive value of FTIRS to diagnose cross transmissions compared to WGS | Month 24
  Positive predictive value
Negative predictive value of FTIRS to diagnose cross transmissions compared to WGS | Month 24
  Negative predictive value

CONTACTS AND LOCATIONS:
Overall Officials: Camille Jeanne-Leroyer, PharmD, Principal Investigator — Caen Normandie Hospital; Olivier Join-Lambert, MD, PhD, Study Director — Caen Normandie University and Hospital
Locations (1):
- CHU CHEN, Caen, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Novais A, Freitas AR, Rodrigues C, Peixe L. Fourier transform infrared spectroscopy: unlocking fundamentals and prospects for bacterial strain typing. Eur J Clin Microbiol Infect Dis. 2019 Mar;38(3):427-448. doi: 10.1007/s10096-018-3431-3. Epub 2018 Nov 27. PMID 30483997
- [Background] Cordovana M, Mauder N, Kostrzewa M, Wille A, Rojak S, Hagen RM, Ambretti S, Pongolini S, Soliani L, Justesen US, Holt HM, Join-Lambert O, Hello SL, Auzou M, Veloo AC, May J, Frickmann H, Dekker D. Classification of Salmonella enterica of the (Para-)Typhoid Fever Group by Fourier-Transform Infrared (FTIR) Spectroscopy. Microorganisms. 2021 Apr 15;9(4):853. doi: 10.3390/microorganisms9040853. PMID 33921159
- [Background] Silva L, Rodrigues C, Lira A, Leao M, Mota M, Lopes P, Novais A, Peixe L. Fourier transform infrared (FT-IR) spectroscopy typing: a real-time analysis of an outbreak by carbapenem-resistant Klebsiella pneumoniae. Eur J Clin Microbiol Infect Dis. 2020 Dec;39(12):2471-2475. doi: 10.1007/s10096-020-03956-y. Epub 2020 Jul 8. PMID 32643025
- [Background] Dinkelacker AG, Vogt S, Oberhettinger P, Mauder N, Rau J, Kostrzewa M, Rossen JWA, Autenrieth IB, Peter S, Liese J. Typing and Species Identification of Clinical Klebsiella Isolates by Fourier Transform Infrared Spectroscopy and Matrix-Assisted Laser Desorption Ionization-Time of Flight Mass Spectrometry. J Clin Microbiol. 2018 Oct 25;56(11):e00843-18. doi: 10.1128/JCM.00843-18. Print 2018 Nov. PMID 30135233
- [Background] Rakovitsky N, Frenk S, Kon H, Schwartz D, Temkin E, Solter E, Paikin S, Cohen R, Schwaber MJ, Carmeli Y, Lellouche J. Fourier Transform Infrared Spectroscopy Is a New Option for Outbreak Investigation: a Retrospective Analysis of an Extended-Spectrum-Beta-Lactamase-Producing Klebsiella pneumoniae Outbreak in a Neonatal Intensive Care Unit. J Clin Microbiol. 2020 Apr 23;58(5):e00098-20. doi: 10.1128/JCM.00098-20. Print 2020 Apr 23. PMID 32161093